CLINICAL TRIAL: NCT01233830
Title: A Phase I, Single Centre, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral AZD2423 Solution After Administration of Multiple Ascending Doses for 12 Days in Young and Elderly Healthy Japanese Volunteers
Brief Title: Study to Investigate Safety, Tolerability and Pharmacokinetics of AZD2423 Multiple Doses in Healthy Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D2600C00004
Record Dates: First submitted 2010-10-19; First posted 2010-11-03 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: safety, tolerability, pharmacokinetics, AZD2423, Japanese

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD2423
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2423 — oral solution
  Arms: 1
Drug: Placebo — oral solution
  Arms: 2

SUMMARY:
The purpose of this study is to assess safety, tolerability and pharmacokinetics of AZD2423 in young and elderly healthy Japanese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy Japanese male volunteers aged ≥20 to ≤45 years and healthy Japanese male and female volunteers aged ≥65 to ≤80 years with suitable veins for cannulation or repeated venipuncture
* Have a body mass index (BMI) between ≥17 and ≤27 kg/m2, as calculated by the investigator(s), and weigh at least 45 kg and no more than 100 kg
* Clinically normal physical findings including supine blood pressure, pulse rate, ECG, and laboratory assessments in relation to age, as judged by the investigator(s)

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator(s), may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically significant illness/infection or medical/surgical procedure or trauma, as judged by the investigator(s), within 3 months of the first administration of investigational product or known malignancy within the past 5 years (with the exception of successfully treated basal cell carcinoma)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse events | Ranging from screening visit (Visit Day 1) to follow-up visit (Visit Day 3)
Vital signs | Ranging from screening visit (Visit Day 1) to follow-up visit (Visit Day 3)
  Changes from baseline in systolic blood pressure, pulse rate and body temperature
Electrocardiograms | Ranging from screening visit (Visit Day 1) to follow-up visit (Visit Day 3)
Laboratory Variables (hematology, urinalysis and clinical chemistry) | Ranging from screening visit (Visit Day 1) to follow-up visit (Visit Day 3)

SECONDARY OUTCOMES:
Plasma concentration over time | Pre-dose, 20 and 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60 and 72 hours after the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Bror Jonzon, MD, PhD, Study Director — AstraZeneca R&D Södertälje; Akimasa Watanabe, Principal Investigator — Kyushu Clinical Pharmacology Research Clinic
Locations (1):
- Research Site, Fukuoka, Japan